CLINICAL TRIAL: NCT05864209
Title: An Intervention to Reduce Phthalate and Bisphenol Exposure During the Critical Period of Minipuberty
Brief Title: Phthalate and Bisphenol Exposure During Minipuberty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-00367
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Phthalate Exposure; Bisphenol Exposure
MeSH Terms: interventions — phthalic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Half of the participants will be randomly assigned to the intervention group and will receive a three-month supply of phthalate- and bisphenol-free baby products (e.g., wipes, diaper cream) and a subscription to a cloth diaper service. Participants will be contacted after 2 and 6 weeks over the phone and administered a brief adherence survey.
  Interventions: Other: Phthalate- and Bisphenol-free Baby Products; Other: Cloth Diapers
- Control Group (Active Comparator): Half of the participants will be randomly assigned to the control group and provided with a three-month supply of conventional disposable diapers (e.g., Huggies or Pampers) and baby products (e.g., wipes, diaper cream). Participants will be contacted after 2 and 6 weeks over the phone and administered a brief adherence survey.
  Interventions: Other: Conventional Disposable Diapers; Other: Conventional Baby Products

INTERVENTIONS:
Other: Phthalate- and Bisphenol-free Baby Products — 3-month supply. Products include wipes and diaper cream.
  Arms: Intervention Group
Other: Cloth Diapers — Subscription to cloth diaper service.
  Arms: Intervention Group
Other: Conventional Disposable Diapers — 3-month supply.
  Arms: Control Group
Other: Conventional Baby Products — Products include wipes and diaper cream.
  Arms: Control Group

SUMMARY:
Phthalates and bisphenols have been detected in a range of infant care products. This pilot study will test whether intervening on these sources of exposure during the critical period of minipuberty affects infants' body burden of phthalates and bisphenols. Investigators will recruit 10 participants from the ongoing NYU Children's Health and Development Study (CHES) cohort study who are >=37 weeks gestation, carrying a male fetus, and intending to breastfeed. Investigators will randomly assign them to use either conventional baby products or phthalate- and bisphenol-free baby products for the first three months of their children's lives. Toward the end of the intervention, investigators will collect maternal breast milk and infant urine, and assay samples for phthalate metabolite and bisphenol concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in NYU CHES study at the NYULH-Brooklyn campus
2. 18 years of age or older
3. At least 37 weeks gestation
4. Carrying a male singleton fetus
5. Intending to breastfeed
6. English or Spanish speaking
7. Intending for pediatric care for infant to occur at the Sunset Park Family Health Center at NYU Langone

Exclusion Criteria:

1. Not enrolled in NYU CHES study from the NYULH-Brooklyn campus
2. Under 37 weeks gestation
3. Carrying a female fetus
4. Carrying multiples
5. Not intending to breastfeed
6. Not comfortable communicating in English or Spanish
7. Not intending for pediatric care for infant to occur at NYULH Sunset Park Family Health Center
8. Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda G Kahn, PhD, MPH, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Sunset Park Family Health Center at NYU Langone - Second Avenue, Brooklyn, New York
  - Tisch Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: linda.kahn@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to linda.kahn@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Infants were not considered enrolled participants for the purpose of this study; infant urine samples were submitted voluntarily by enrolled (mother) participants at home during follow-up. Participant information (participant flow, baseline characteristics) are thus not reported for infants.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 5 | 5
Completed | 3 | 2
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.02 (3.96) | 33.025 (13.20) | 30.023 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Log Signal Intensity of Bisphenol A (BPA) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via non-targeted HPLC-MS/MS. The log signal intensity, an arbitrary unit, is a measurement of the signal strength of BPA in child urine; as the concentration of BPA increases, the signal intensity increases proportionally in a logarithmic fashion; higher values indicate greater infant exposure to bisphenol.
Time Frame: Month 3
Population: 3 out of 5 participants in the intervention group and 2 out of 5 in the control group were analyzed as the rest did not provide samples
Measure: Mean (Standard Deviation); unit: Log(Arbitrary Units)
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 3 | 2
Log(Arbitrary Units) | 0.00 (0.00) | 5.43 (0.16)

2. Primary Outcome: Log Signal Intensity of Bisphenol A (BPA) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via non-targeted HPLC-MS/MS. The log signal intensity, an arbitrary unit, is a measurement of the signal strength of BPA in child urine; as the concentration of BPA increases, the signal intensity increases proportionally in a logarithmic fashion; higher values indicate greater maternal exposure to bisphenol.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Log(Arbitrary Units)
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 3 | 2
Log(Arbitrary Units) | 3.49 (2.47) | 4.74 (0.40)

3. Secondary Outcome: Mean Concentrations of Monomethyl Phthalate (mMP) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: Only one intervention and one control sample was collected for child urine
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 1 | 1
microgram/gram creatinine | 27.23 (NA) — n=1 participant analyzed. | 13.79 (NA) — n=1 participant analyzed.

4. Secondary Outcome: Mean Concentrations of Monomethyl Phthalate (mMP) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: 3 out of 5 participants in the intervention group anf 2 out of 5 in the control group were analyzed as the rest did not provide samples
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 3 | 2
microgram/gram creatinine | 2.91 (2.66) | 5.10 (0.41)

5. Secondary Outcome: Mean Concentrations of Monoethyl Phthalate (mEP) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: Only one intervention and one control sample was collected for child urine
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 1 | 1
microgram/gram creatinine | 129.68 (NA) — N=1 participant analyzed. | 1649.72 (NA) — N=1 participant analyzed.

6. Secondary Outcome: Mean Concentrations of Monoethyl Phthalate (mEP) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 3 | 2
microgram/gram creatinine | 89.40 (74.36) | 53.30 (8.78)

7. Secondary Outcome: Mean Concentrations of Phthalic Acid (PA) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: Only one intervention and one control sample was collected for child urine
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 1 | 1
microgram/gram creatinine | 24.18 (NA) — N=1 Participant analyzed. | 161.58 (NA) — N=1 Participant analyzed.

8. Secondary Outcome: Mean Concentrations of Phthalic Acid (PA) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 3 | 2
microgram/gram creatinine | 63.96 (91.12) | 211.21 (126.69)

9. Secondary Outcome: Mean Concentrations of Mono-(2-ethyl-5-hydroxyhexyl) Phthalate (mEHHP) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: Only one intervention and one control sample was collected for child urine
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 1 | 1
microgram/gram creatinine | 0.42 (NA) — N=1 participant analyzed. | 6.81 (NA) — N=1 participant analyzed.

10. Secondary Outcome: Mean Concentrations of Mono-(2-ethyl-5-hydroxyhexyl) Phthalate (mEHHP) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 3 | 5
microgram/gram creatinine | 8.15 (7.19) | 2.43 (0.98)

11. Secondary Outcome: Mean Concentrations of Mono-carboxy-isooctyl Phthalate (mCIOP) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 1 | 1
microgram/gram creatinine | 0.50 (NA) — N=1 participant analyzed | 2.92 (NA) — N=1 participant analyzed

12. Secondary Outcome: Mean Concentrations of Mono-carboxy-isooctyl Phthalate (mCIOP) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 3 | 2
microgram/gram creatinine | 1.90 (1.25) | 2.12 (1.08)

13. Secondary Outcome: Mean Concentrations of Monobutyl Phthalate (mBP) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: Only one intervention and one control sample was collected for child urine.
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 1 | 1
microgram/gram creatinine | 62.77 (NA) — N=1 participant analyzed | 37.40 (NA) — N=1 participant analyzed

14. Secondary Outcome: Mean Concentrations of Monobutyl Phthalate (mBP) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 3 | 2
microgram/gram creatinine | 18.02 (7.21) | 21.75 (19.88)

15. Secondary Outcome: Mean Concentrations of Mono-iso-butyl Phthalate (mIBP) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: Only one intervention and one control sample was collected for child urine
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 1 | 1
microgram/gram creatinine | 74.45 (NA) — N=1 participant analyzed | 28.25 (NA) — N=1 participant analyzed

16. Secondary Outcome: Mean Concentrations of Mono-iso-butyl Phthalate (mIBP) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 3 | 2
microgram/gram creatinine | 13.07 (10.02) | 10.12 (7.04)

17. Secondary Outcome: Mean Concentrations of Mono(5-carboxy-2-ethylpentyl) Phthalate (mECPP) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: Only one intervention and one control sample was collected for child urine
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 1 | 1
microgram/gram creatinine | 2.51 (NA) — N=1 participant analyzed | 20.00 (NA) — N=1 participant analyzed

18. Secondary Outcome: Mean Concentrations of Mono(5-carboxy-2-ethylpentyl) Phthalate (mECPP) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 3 | 2
microgram/gram creatinine | 8.27 (6.6) | 3.06 (0.58)

19. Secondary Outcome: Mean Concentrations of Mono-(2-ethyl-5-oxohexyl) Phthalate (mEOHP) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: Only one intervention and one control sample was collected for child urine
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 1 | 1
microgram/gram creatinine | 0.39 (NA) — N=1 participant analyzed | 5.06 (NA) — N=1 participant analyzed

20. Secondary Outcome: Mean Concentrations of Mono-(2-ethyl-5-oxohexyl) Phthalate (mEOHP) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 3 | 2
microgram/gram creatinine | 4.34 (3.16) | 1.37 (0.49)

21. Secondary Outcome: Mean Concentrations of Bisphenol S (BPS) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: Only one intervention and one control sample was collected for child urine
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 1 | 1
microgram/gram creatinine | 2.09 (NA) — N=1 participant analyzed | 1.61 (NA) — N=1 participant analyzed

22. Secondary Outcome: Mean Concentrations of Bisphenol S (BPS) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: 2 out of 5 participants in the intervention group and 2 out of 5 in the control group were analyzed as the rest did not provide samples
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 2 | 2
microgram/gram creatinine | 1.80 (0.82) | 0.57 (0.58)

23. Secondary Outcome: Mean Concentrations of Mono-carboxy-isononyl Phthalate (mCINP) in Maternal Urine Samples
Description: Maternal urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 2 | 2
microgram/gram creatinine | 0.59 (0.31) | 1.52 (1.92)

24. Secondary Outcome: Mean Concentrations of Ono-carboxy-isononyl Phthalate (mCINP) in Child Urine Samples
Description: Child urine samples were analyzed for bisphenols and for phthalate metabolites via targeted LC-MS/MS.
Time Frame: Month 3
Population: Only one intervention and one control sample was collected for child urine
Measure: Mean (Standard Deviation); unit: microgram/gram creatinine
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 1 | 1
microgram/gram creatinine | 0.61 (NA) — N=1 participant analyzed. | 1.06 (NA) — N=1 participant analyzed.

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT05864209/Prot_SAP_000.pdf